CLINICAL TRIAL: NCT06865807
Title: Influence of Suture Type on Emergency Midline Laparotomy Closure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital San Juan de Dios Tenerife (Other)
Responsible Party: Principal Investigator, Julen Ramon Rodríguez, Principal Investigator, University Hospital of the Nuestra Señora de Candelaria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 52/24
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Linea Alba Hernia; Evisceration; Operation Wound; Suture; Complications, Mechanical

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PDS (Active Comparator): Closure emergency laparotomy using PDS 2/0 small bites
  Interventions: Procedure: PDS 2/0 vs Monomax 2/0
- Monomax (Experimental): Closure emergency laparotomy using Monomax 2/0 small bites
  Interventions: Procedure: PDS 2/0 vs Monomax 2/0

INTERVENTIONS:
Procedure: PDS 2/0 vs Monomax 2/0 — We will include in the study patients who require an emergency midline laparotomy by the General and Digestive Surgery Department of the University Hospital Nuestra Señora de Candelaria. Patients will be randomized based on their medical record number: those with an even number will undergo laparotomy closure using PDS 2/0, and those with an odd number will receive Monomax 2/0.

SUMMARY:
There is no clear recommendation in international guidelines regarding the type of suture to be used for closing emergency midline laparotomies. It is recommended to follow the same principles as in elective surgery, thus performing the closure with a continuous suture of slowly absorbable monofilament 2-0 with small-bites technique. Currently, there are several slowly absorbable sutures available on the market, and our center uses two: PDS® and Monomax®. These two sutures are currently used interchangeably at our institution based on the preferences of each surgeon.

Objective: study whether there are differences between these two sutures in the closure of emergency midline laparotomy.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old, patients undergoing emergency midline laparotomy by the General Surgery Department.

Exclusion Criteria:

* <18 years old, previous midline laparotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-12-10 (Estimated)

PRIMARY OUTCOMES:
Evisceration | 1 month
  Rate of evisceration

SECONDARY OUTCOMES:
Wound complication | 1 month
  Seroma, hematoma, infection
Incisional hernia | 1 year
  Evaluate the rate of incisional hernia during follow-up in outpatient consultations.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Nuestra Señora de Candelaria, Santa Cruz de Tenerife, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bosanquet DC, Ansell J, Abdelrahman T, Cornish J, Harries R, Stimpson A, Davies L, Glasbey JC, Frewer KA, Frewer NC, Russell D, Russell I, Torkington J. Systematic Review and Meta-Regression of Factors Affecting Midline Incisional Hernia Rates: Analysis of 14,618 Patients. PLoS One. 2015 Sep 21;10(9):e0138745. doi: 10.1371/journal.pone.0138745. eCollection 2015. PMID 26389785
- [Background] Muysoms FE, Antoniou SA, Bury K, Campanelli G, Conze J, Cuccurullo D, de Beaux AC, Deerenberg EB, East B, Fortelny RH, Gillion JF, Henriksen NA, Israelsson L, Jairam A, Janes A, Jeekel J, Lopez-Cano M, Miserez M, Morales-Conde S, Sanders DL, Simons MP, Smietanski M, Venclauskas L, Berrevoet F; European Hernia Society. European Hernia Society guidelines on the closure of abdominal wall incisions. Hernia. 2015 Feb;19(1):1-24. doi: 10.1007/s10029-014-1342-5. Epub 2015 Jan 25. PMID 25618025
- [Background] Frassini S, Cobianchi L, Fugazzola P, Biffl WL, Coccolini F, Damaskos D, Moore EE, Kluger Y, Ceresoli M, Coimbra R, Davies J, Kirkpatrick A, Di Carlo I, Hardcastle TC, Isik A, Chiarugi M, Gurusamy K, Maier RV, Segovia Lohse HA, Jeekel H, Boermeester MA, Abu-Zidan F, Inaba K, Weber DG, Augustin G, Bonavina L, Velmahos G, Sartelli M, Di Saverio S, Ten Broek RPG, Granieri S, Dal Mas F, Fare CN, Peverada J, Zanghi S, Vigano J, Tomasoni M, Dominioni T, Cicuttin E, Hecker A, Tebala GD, Galante JM, Wani I, Khokha V, Sugrue M, Scalea TM, Tan E, Malangoni MA, Pararas N, Podda M, De Simone B, Ivatury R, Cui Y, Kashuk J, Peitzman A, Kim F, Pikoulis E, Sganga G, Chiara O, Kelly MD, Marzi I, Picetti E, Agnoletti V, De'Angelis N, Campanelli G, de Moya M, Litvin A, Martinez-Perez A, Sall I, Rizoli S, Tomadze G, Sakakushev B, Stahel PF, Civil I, Shelat V, Costa D, Chichom-Mefire A, Latifi R, Chirica M, Amico F, Pardhan A, Seenarain V, Boyapati N, Hatz B, Ackermann T, Abeyasundara S, Fenton L, Plani F, Sarvepalli R, Rouhbakhshfar O, Caleo P, Ho-Ching Yau V, Clement K, Christou E, Castillo AMG, Gosal PKS, Balasubramaniam S, Hsu J, Banphawatanarak K, Pisano M, Adriana T, Michele A, Cioffi SPB, Spota A, Catena F, Ansaloni L. ECLAPTE: Effective Closure of LAParoTomy in Emergency-2023 World Society of Emergency Surgery guidelines for the closure of laparotomy in emergency settings. World J Emerg Surg. 2023 Jul 26;18(1):42. doi: 10.1186/s13017-023-00511-w. PMID 37496068
- [Background] Thorup T, Tolstrup MB, Gogenur I. Reduced rate of incisional hernia after standardized fascial closure in emergency laparotomy. Hernia. 2019 Apr;23(2):341-346. doi: 10.1007/s10029-019-01893-0. Epub 2019 Jan 25. PMID 30684103